CLINICAL TRIAL: NCT07118709
Title: A Phase I Study to Evaluate the Safety,Tolerability, Pharmacokinetics and Preliminary Efficacy of KC1086 in the Patients With Advanced Recurrent or Metastatic Solid Tumors
Brief Title: A Study of KC1086 in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Konruns Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KC1086-I-01
Record Dates: First submitted 2025-08-01; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KC1086 (Experimental): KC1086 are given orally once daily, 21 days as a cycle
  Interventions: Drug: KC1086

INTERVENTIONS:
Drug: KC1086 — Part 1: Dose-escalation phase , five dose groups are included: 1 mg, 2 mg, 4 mg, 6 mg, and 8 mg.
  Part 2: Dose-expansion phase, 2 to 3 dose levels will be selected for expansion based on the results of the dose escalation phase.

SUMMARY:
The purpose of this study is to evaluate the safety，tolerability, pharmacokinetics, and preliminary efficacy of KC1086 in participants with advanced recurrent or metastatic solid tumors. The trial will be divided into two parts: dose-escalation phase and dose-expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed recurrent or metastatic solid tumors;
2. Patients who have failed standard or conventional treatment or for whom no standard treatment is available( definition of treatment failure: intolerable toxic and side effects, disease progression during treatment recurrence after treatment);
3. Participants with advanced recurrent, unresectable, and/or metastatic tumors must have evaluable or measurable lesions (according to RECIST 1.1)；
4. Eastern Cooperative Oncology Group performance status score of 0 or 1;
5. Life expectancy > 12 weeks;
6. Adequate bone marrow, renal, and hepatic function;
7. Patients should participate in the study voluntarily and sign informed consent.

Exclusion Criteria:

1. Any patient who is known to have untreated central nervous system (CNS) metastasis;
2. Other kinds of malignancies within 5 years;
3. Gastrointestinal abnormalities;
4. Cardiovascular and cerebrovascular diseases;
5. Involved in other clinical trials within 4 weeks before enrollment;
6. Prior anti-tumor therapies with radiotherapy, immunotherapy, operation within 4 weeks before enrollment;
7. Prior anti-tumor therapies with small molecule targeting drugs within 2weeks or 5 half-lives (whichever is longer) before enrollment; Prior anti-tumor therapies with chemotherapy within 3 weeks or 5 half-lives (whichever is longer) before enrollment;
8. Presence of unresolved toxicities from prior anti-tumor therapy, defined as having not resolved to NCI CTCAE 5.0 Grade 0 or 1;
9. Severe infection within 4 weeks prior to enrollment;
10. Uncontrolled massive ascites, pleural or pericardial effusion；
11. Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy;
12. Prior therapies with KAT6 inhibitors
13. Pregnant or lactating women;
14. Female subjects of child-bearing potential and male subjects of reproductive capacity who do not agree to use contraceptive measures during the study and for 6 months after the end of the study.
15. Other patients are not eligible for enrollment assessed by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | approximately 3 years
  Incidence of treatment-related AEs

SECONDARY OUTCOMES:
Pharmacokinetics (PK) profile: Cmax | approximately 3 years
  Peak Plasma Concentration
Pharmacokinetics (PK) profile: Tmax | approximately 3 years
  Time to reach the maximum plasma concentration
Pharmacokinetics (PK) profile: T1/2 | approximately 3 years
  Terminal half-life
Pharmacokinetics (PK) profile: AUC0-t and AUC0-∞ | approximately 3 years
  Area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration, or Area under the single-dose plasma concentration-time curve from Hour 0 to infinity
Objective Response Rate (ORR) | approximately 3 years
  Overall response rate (ORR) was defined as the percentage of participants with a best overall complete response (CR) or partial response (PR) per RECIST 1.1.
Progression-free survival (PFS) | approximately 3 years
  Progression-free survival (PFS) was defined as the time from the start date of study drug to the date of the first radiologically documented progressive disease (PD) per RECIST 1.1 or death due to any cause.
Disease Control Rate (DCR) | approximately 3 years
  Disease Control Rate (DCR) was defined as the percentage of participants with a best overall complete response (CR), partial response (PR), or stable disease (SD) per RECIST 1.1.
Duration of Response (DOR) | approximately 3 years
  Duration of response (DOR) was defined as the time from first documented response (partial response (PR) or complete response (CR)) to the date of first documented disease progression (PD) or death due to any cause, among patients with a confirmed PR or CR per RECIST 1.1.

IPD SHARING:
Plan to Share IPD: No